CLINICAL TRIAL: NCT00030823
Title: Vaccination Of High Risk Breast Cancer Patients With Heptavalent Antigen - Keyhole Limpet Hemocyanin Conjugate Plus The Immunological Adjuvant QS21
Brief Title: Vaccine Therapy in Treating Patients at High Risk for Breast Cancer Recurrence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-019; MSKCC-01019; NCI-H01-0084
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Results first posted 2015-12-30 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — saponin QA-21V1

ARMS (1):
- Vaccine (Experimental): Patients receive Globo-H-GM2-Lewis-y-MUC1-32(aa)-sTn(c)-TF(c)-Tn(c)-KLH conjugate vaccine with QS21 adjuvant subcutaneously weekly on weeks 1, 2, 3, 7, and 19.
  Interventions: Biological: Globo-H-GM2-Lewis-y-MUC1-32(aa)-sTn(c)-TF(c)-Tn(c)-KLH conjugate vaccine; Biological: QS21

INTERVENTIONS:
Biological: Globo-H-GM2-Lewis-y-MUC1-32(aa)-sTn(c)-TF(c)-Tn(c)-KLH conjugate vaccine
Biological: QS21

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response and decrease the recurrence of breast cancer.

PURPOSE: Pilot trial to study the effectiveness of vaccine therapy in treating patients who are at high risk for breast cancer recurrence.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether immunization with multiple antigens comprising GM2, Globo-H, Lewis y, TF(c), sTn(c), Tn(c), and glycosylated MUC-1 32(aa) conjugated to keyhole limpet hemocyanin plus QS21 induces an antibody response against these individual antigens and breast cancer cells expressing these antigens in patients at high risk for breast cancer recurrence.
* Determine the toxic effects of this regimen in these patients.

OUTLINE: Patients receive Globo-H-GM2-Lewis-y-MUC1-32(aa)-sTn(c)-TF(c)-Tn(c)-KLH conjugate vaccine with QS21 adjuvant subcutaneously weekly on weeks 1, 2, 3, 7, and 19.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 2-3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer at high risk for recurrence, defined by one of the following:

  * Stage IV that is free of all known disease after eradication by surgery, radiotherapy, or chemotherapy

    * May or may not have elevated CA 15-3 or CEA levels
  * Stage I, II, or III previously treated with adjuvant chemotherapy and clinically free of identifiable disease, but have rising CA 15-3 or CEA levels

    * Rising CA 15-3 and CEA defined as a prior normal level increased on 2 consecutive occasions at least 2 weeks apart

      * For patients with a significant history of smoking who have a chronically elevated CEA (less than 15), CEA must be increased at least 1.5 times the uppermost chronic value on 2 consecutive occasions at least 2 weeks apart
  * Stage III and completed adjuvant therapy no more than 24 months ago
  * Recurrence in the ipsilateral axilla after lumpectomy and/or axillary dissection or modified radical mastectomy
  * Recurrence in the ipsilateral breast after lumpectomy and/or axillary dissection
  * Stage II with at least 4 positive axillary nodes and completed adjuvant therapy no more than 24 months ago
  * Stage IV that is stable on hormonal therapy
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Male or female

Menopausal status:

* Not specified

Performance status:

* Karnofsky 80-100%

Life expectancy:

* Not specified

Hematopoietic:

* Lymphocyte count at least 500/mm^3
* WBC at least 3,000/mm^3

Hepatic:

* AST no greater than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 1.5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No clinically significant New York Heart Association class III or IV cardiac disease

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior seafood allergy
* No known prior immunodeficiency or autoimmune disease
* No other active cancer except basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 6 weeks since prior immunotherapy
* No prior vaccine with any of the antigens in this study

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* At least 4 weeks since prior surgery
* Concurrent surgery for local recurrence allowed if patient remains disease free

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2001-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Ann Gilewski, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Armstrong JL, Ragupathi G, Powell S, et al.: Preliminary data of vaccination of high risk breast cancer (BC) patients (pts) with a heptavalent antigen: keyhole limpet hemocyanin (KLH) conjugate plus the immunologic adjuvant QS-21. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-675, 2003.
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vaccine
Started | 14
Completed | 13
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vaccine
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety
Description: By assessing the toxicity and will be graded following immunization with polyvalent vaccine in accordance with the NCI Common Toxicity Criteria 2.0.
Time Frame: 2 years
Population: All 13 participants experienced toxicities.
Measure: Number; unit: participants
Arm/Group | Vaccine
Number analyzed (Participants) | 13
participants | 13

ADVERSE EVENTS:
Arm/Group | Vaccine
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine (N=13)
SGPT (ALT) (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine (N=13)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 2 (4)
Derm, skin other (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspepsia/heartburn (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 4 (7)
Fever (General disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Injection site reaction (Infections and infestations) | 13 (39)
Leukocytes (Blood and lymphatic system disorders) | 1 (1)
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, other (General disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2)
Rigors, chills (General disorders) | 1 (1)
SGOT (AST) (Blood and lymphatic system disorders) | 1 (2)
SGPT (ALT) (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes